CLINICAL TRIAL: NCT01941511
Title: A Phase 1, Randomized, 3-way, Crossover Single Dose, Placebo, and Active Controlled Study to Evaluate the Effect of Intravenous Doses of GMI-1070 on Qtc Intervals in Healthy African-American Adult Subjects
Brief Title: A Study to Evaluate the Effect of IV Doses of GMI-1070 on Qtc Intervals in Healthy African-American Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: B5201001; B5201001
Record Dates: First submitted 2013-08-27; First posted 2013-09-13 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: QTc; African-American; GMI-1070; QT/QTc interval prolongation
MeSH Terms: interventions — rivipansel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rivipansel/Placebo/Moxifloxacin (Experimental): Rivipansel 4.8 gA IV infusion over 20 minutes Phosphate Buffered Saline (PBS) IV infusion over 20 minutes Moxifloxacin (Avelox) 400 mg single oral dose
  Interventions: Drug: Rivipansel

INTERVENTIONS:
Drug: Rivipansel — Subjects will receive in a randomized sequence rivipansel 4gA IV, moxifloxacin 400 mg, and placebo IV.
  Other Names: GMI-1070

SUMMARY:
This is a clinical evaluation of QT/QTc interval prolongation and proarrhythmic potential of GMI-1070 in African-American Adult subjects. This is conducted as part of standard drug development.

DETAILED DESCRIPTION:
Safety

ELIGIBILITY:
Inclusion Criteria:

* Healthy African-American male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive.

Exclusion Criteria:

* Pregnant females; breastfeeding females; and females of childbearing potential. Males who are unwilling or unable to use 2 highly effective method of contraception for the duration of the study starting at least 14 days prior to the first dose of investigational product and for at least 28 days after the last dose of investigational product.
* Non African-American.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic,seasonal allergies at the time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
QTc, during rivipansel treatment period | prior to dose, through 72 hours after dosing
  QTc, using Fridericia's correction method (QTcF) at each time point during rivipansel treatment period.
QTc, during placebo treatment period | prior to dose, through 72 hours after dosing
  QTc, using Fridericia's correction method (QTcF) at each time point during placebo treatment period.

SECONDARY OUTCOMES:
QTc, during moxifloxacin treatment period | prior to dose, through 72 hours after dosing
  QTcF, or any other appropriate correction method at each postdose time point of moxifloxacin treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, San Antonio, Texas, United States